CLINICAL TRIAL: NCT04788615
Title: Open-Label Rater-Blind Randomized Multi-Center Parallel-Arm Active- Comparator Study to Assess the Efficacy and Tolerability of Ofatumumab 20mg SC Monthly vs. First Line DMT - Physician's Choice in the Treatment of Newly Diagnosed RMS
Brief Title: Open Label Randomized Multicenter to Assess Efficacy & Tolerability of Ofatumumab 20mg vs. First Line DMT in RMS
Acronym: STHENOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COMB157G3301; 2020-004505-32 (EudraCT Number)
Record Dates: First submitted 2021-03-08; First posted 2021-03-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
Keywords: Ofatumumab; relapsing multiple sclerosis; relapsing-remitting MS; MS therapy; RMS; Relapsing MS; Glatiramer acetate; IFNβ-1b; IFNβ-1a; peg-IFNβ-1a; Teriflunomide; Dimethyl fumarate; Diroximel fumarate; OMB157; adult
MeSH Terms: conditions — Multiple Sclerosis | interventions — ofatumumab; Glatiramer Acetate; Interferons; teriflunomide; Dimethyl Fumarate; diroximel fumarate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The independent EDSS (Expanded disability status scale) rater will be blind to the identity of the treatment throughout the study period. Patient MRI scans read by an independent central MRI reading center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ofatumumab (Experimental): Oftatumumab 20mg auto injector syringes for subcutaneous injection on Day 1, Week 1 and 2, followed by subsequent monthly dosing, starting at Month 1.
  Interventions: Drug: Ofatumumab
- First line DMT (Active Comparator): 1. Glatiramer acetate minimum dose 20mg or maximum dose 40mg twice a day or three times a week or
  2. Interferon minimum dose 22µg or maximum dose of 0.25mg 3 times a week or once a week or Every second week depending on preparation or
  3. Peg-Interferon beta-1a minimum dose of 63µg or maximum dose of 125µg every 2 weeks (14 days) or
  4. Teriflunomide 14 mg once a day or
  5. Dimethyl fumarate minimum dose of 120mg or maximum dose of 240mg twice a day
  6. Diroximel fumarate minimum dose of 231mg or maximum dose of 462mg twice a day
  Interventions: Drug: First line DMT

INTERVENTIONS:
Drug: Ofatumumab — 20mg Subcutaneous injection
  Other Names: OMB157
  Arms: ofatumumab
Drug: First line DMT — any one of these based on availability at country given as First line DMT Glatiramer acetate 20mg or 40mg or Interferon 22µg or 0.25mg or Peg-Interferon beta-1a 63µg or 125µg or Teriflunomide 14mg or Dimethyl fumarate 120mg or 240mg or Diroximel fumarate 231mg or 462mg
  Other Names: Glatiramer acetate or Interferon or Peg-Interferon beta-1a or Teriflunomide or Dimethyl fumarate or Diroximel fumarate
  Arms: First line DMT

SUMMARY:
This study will compare ofatumumab vs. European approved platform first line self-administered disease modifying therapy (DMT) in newly diagnosed MS patients

DETAILED DESCRIPTION:
The study is a randomized (1:1), open-label, rater-blind, multi-center, prospective, parallel-arm, active comparator study which will consist of 15 months treatment period and a 6 months observational safety extension period, for patients who withdraw ofatumumab for any reason, in 186 total patients with early relapsing multiple sclerosis (RMS) RMS patients are patients who are newly diagnosed or have never been on active treatment at the time of study entry with ≤ 5 years from first MS symptoms.

There is a screening period and patients are randomized to either ofatumumab or first line DMT at baseline. Patients will be treated until the end of study (EOS) or for a maximum duration of 15 months. Patients who prematurely discontinue study drug or comparator will have their end of treatment (EOT) visit and assessments at the time of discontinuation. After ofatumumab or the standard of care comparator (DMT) discontinuation, patients may initiate alternative MS therapy according to local standard of care, if clinically indicated.

Patients who for any reason withdraw from ofatumumab during treatment will be invited to participate in the observational extension safety period for 6 months or until patient re-starts MS treatment with a new DMT treatment. During this period, clinical efficacy after ofatumumab withdrawal will be assessed.

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent obtained before any assessment
2. Male/female patients, 18 through 55 (inclusive) years of age.
3. Diagnosis of MS according to the 2017 revised McDonald criteria (Thompson et al 2018).
4. Relapsing MS: relapsing-course (RMS), as defined by Lublin et al 2014.
5. Treatment Naïve patients, ≤ 5 years since first MS symptom.
6. EDSS score 0-4.0 (inclusive).
7. Patient must be suitable to be treated with one of first line self-administered DMT-physician's choice (glatiramer acetate, IFNs, teriflunomide, DMF, diroximel fumarate according to EMA SmPC) or ofatumumab depending on randomization and physician's choice
8. At least 1 relapse or 1 Gd+ enhanced lesion on T1 in 1 year prior to Screening.
9. Able to obtain MRI assessment.
10. Neurologically stable within 1 month prior to first study drug administration Exclusion Criteria

<!-- -->

1. Diseases other than multiple sclerosis responsible for the clinical or MRI presentation
2. Progressive MS phenotypes: Patients with primary progressive MS (Polman et al 2011) or SPMS (Lublin et al 2014).
3. Use of other experimental or investigational drugs at the time of enrollment (Screening) or within the prior 30 days, or 5 elimination half-lives, or until the expected pharmacodynamics effect has returned to baseline, whichever is longer
4. Relapse between Screening and Baseline visits
5. Pregnancy or breastfeeding
6. Patients suspected of not being able or willing to cooperate or comply with study protocol requirements in the opinion of the Investigator
7. Women of childbearing potential defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception (methods that result in less than 1% pregnancy rates) while receiving ofatumumab and for 6 months after the last administration. The requirements for contraception for the comparators should also be taken into consideration according to their SmPC.

   Highly effective methods of contraception include:
   * Total abstinence (when this is in line with the preferred and usual lifestyle of the participant). Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant. Periodic abstinence (e.g. calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.
   * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
   * Male sterilization (at least 6 months prior to screening). For female participants on the study, the vasectomized male partner should be the sole partner for that participant.

   (Vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the WOCBP trial participant and that the vasectomized partner has received medical assessment of the surgical success.) - Use of combined, estrogen and progesterone containing (oral, intravaginal, transdermal), hormonal methods of contraception or use of progesterone-only (oral, injectable, implantable) hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment. Women are considered post-menopausal if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate history of vasomotor symptoms). Women are considered not of childbearing potential if they are post-menopausal or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of childbearing potential. If local regulations deviate from the contraception methods listed above to prevent pregnancy, local regulations apply and will be described in the ICF.
8. Patients with an active chronic disease (or stable but treated with immune therapy) of the immune system other than MS (e.g. rheumatoid arthritis, scleroderma, Sjögren's syndrome, Crohn's disease, ulcerative colitis, etc.) or with immunodeficiency syndrome (hereditary immune deficiency, drug-induced immune deficiency)
9. Patients with an active infection (bacterial, fungal, or viral like hepatitis, HIV or COVID), until the infection is resolved. Where local regulation requires it, Sars-Cov-19 must be ruled out by the PCR test.
10. Patients with neurological findings consistent with Progressive Multifocal Leukoencephalopathy (PML), or confirmed PML
11. Positive results at Screening for serological markers for hepatitis (H) B and C indicating acute or chronic infection:

    - Hepatitis B virus (HBV) screening should be performed before initiation of treatment.

    At a minimum, screening should include hepatitis B surface antigen (HBsAg) and hepatitis B core antibody (HBcAb) testing. These can be complemented with other appropriate markers as per local guidelines. Patients with positive hepatitis B serology (either HBsAg or HBcAb) should consult a liver disease expert before the start of treatment and should be monitored and managed following local medical standards to prevent hepatitis B reactivation.

    - Hepatitis C risk must be ruled out via anti-HC IgG (if positive IgG, HCV-RNA PCR will be performed and if negative, patient can be enrolled) NOTE: If the Investigator suspects false positive hepatitis serology results such as an antibody pattern indicating acute hepatitis infection but no corresponding elevated liver enzymes and no signs or symptoms of liver disease, an infectious disease expert may be consulted. In the case the patient has a record of vaccination including HB, and there is no evidence of acute or chronic hepatitis infection (confirmed by an infectious disease expert), the Investigator must document (in source data and as a comment in the electronic Case Report Form (eCRF) that the serology results are considered false positive and may then enroll the subject.
12. Have received any live or live-attenuated vaccines within 4 weeks prior to first study drug administration
13. Any other disease or condition that could interfere with participation in the study according to the study protocol, or with the ability of the patients to cooperate or comply with the study procedures
14. Any of the following conditions or treatments that may impact the safety of the patient:

    - History of, or current, significant cardiac disease including cardiac failure (NYHA functional class II-IV), myocardial infarction (within 6 months prior to screening), unstable angina (within 6 months prior to screening), transient ischemic attack (within 6 months prior to screening), stroke, cardiac arrhythmias requiring treatment or uncontrolled arterial hypertension

    - Concomitant clinically significant cardiac arrhythmias, e.g. sustained ventricular tachycardia and clinically significant second or third degree AV block without a pacemaker on screening electrocardiogram (ECG)
    * History of or active severe respiratory disease, including Chronic Obstructive Pulmonary Disease, interstitial lung disease or pulmonary fibrosis
    * Patients with asthma requiring regular treatment with oral steroids
    * Severe hepatic impairment (Child-Pugh class C) or any chronic liver or biliary disease
    * Patients with severe renal impairment (glomerular filtration rate < 30 ml/min/1.73 m2)
    * Any medically unstable condition as determined by the Investigator
15. Any of the following abnormal laboratory values prior to first study drug administration:

    - Total bilirubin greater than 3 times upper limit of normal (ULN) range, unless in the context of Gilbert's syndrome

    - Alkaline phosphatase (ALP) greater than 5 times the ULN range

    - Serum IgG < 500mg/dL (according to central laboratory range)
    * Any other clinically significant laboratory assessment as determined by the Investigator (e.g. significant anemia, neutropenia, thrombocytopenia, signs of impaired bone marrow function)
16. Patients with severe hypoproteinemia e.g. in nephrotic syndrome
17. Patients with any of the following neurologic/psychiatric disorders prior to first study drug administration: - Score "yes" on item 4 or item 5 of the Suicidal Ideation section of the Columbia- Suicide Severity Rating Scale (CSSRS) if this ideation occurred in the past 6 months OR

    * "yes" on any item of the Suicidal Behavior section, except for the "Non-Suicidal Self- Injurious Behavior" (item also included in the Suicidal Behavior section) if this behavior occurred in the past 2 years.
18. History of hypersensitivity to the study drug or any of the excipients or to drugs of similar chemical classes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with no evidence of disease activity (NEDA-3) | Baseline to 15 month
  NEDA-3 (yes/no) is defined as:
  1. Absence of confirmed clinical relapse
  2. Absence of new MRI activity (Gd+ T1 lesion or new/enlarged T2 lesion) with MRI re-baselined at Month 3
  3. Absence of 3-month confirmed disability worsening

SECONDARY OUTCOMES:
Number of relapses | Baseline to Month 15
  Number of relapses will be summarized descriptively
Annual relapse rate | Baseline to Month 15
  Annual relapse rate will be analyzed by treatment group using negative binomial regression model with log-link and patient's time in study will be used as an offset.
Percentage of relapse-free patients and proportion of relapse free patients with MRI activity free | Month 3, Month 9 and Month 15
  Proportion of relapse-free patients and proportion of relapse-free patients with MRI activity free at Month 3, 9 and 15 will be summarized descriptively at each timepoint.
Time to 3 month Confirmed Disability Worsening (CDW) and time to 6-month Confirmed Disability Worsening (CDW) | Baseline to Month 3 and to Month 6
  Time to 3 month Confirmed Disability Worsening (CDW) and time to 6-month CDW will be assessed by EDSS (Expanded disability status scale) score
Change in expanded disability status scale (EDSS) | Baseline to Month 15
  Change in expanded disability status scale (EDSS) from baseline to end of study will be summarized descriptively based on the expanded disability status scale (EDSS) score
Percentage of disability-progression free patients | Baseline to Month 15
  Proportion of disability-progression free patients at end of study will be summarized descriptively
Number of Gd+ T1 lesions of brain | Baseline to Month 15
  Number of Gd+ T1 lesions of brain will be summarized descriptively.
The number and percentage of patients with Treatment emergent adverse events (TEAE) or adverse events reports | Baseline to Month 15 and 6 months safety follow-up
  Adverse will be collected at each patients visit including any clinically significant safety assessments determined to be an adverse event by the investigator
Volume of Gd+ T1 lesions of brain | Baseline to Month 15
  Volume of Gd+ T1 lesions of brain will be summarized descriptively.
Number of new/enlarging T2 lesions of brain | Baseline to Month 15
  Number of new/enlarging T2 lesions of brain will be summarized descriptively.
Volume of new enlarging T2 lesions of brain | Baseline to Month 15
  Volume of new enlarging T2 lesions of brain will be summarized descriptively.
Mean time to first relapse | Baseline to Month 15
  Mean time to first relapse will be summarized descriptively
Percentage of SAEs, and SAEs with hospitalizations | Baseline to Month 15 and 6 months safety follow-up
  Proportion of SAEs, and SAEs with hospitalizations between ofatumumab 20 mg s.c. and first line self-administered DMTs
Percentage of treatment compliance of participants | Baseline to Month 15
  Treatment compliance will be assessed by review of participant diary entries and counts of treatment (dispensed and returned)
Percentage of patient with AEs | Baseline to Month 15 and 6 months safety follow-up
  Proportion of patients with adverse events, including injection related reactions
Percentage of withdrawn patients | Baseline to Month 15
  Proportion of patients who withdrew due to abnormal lab values
Percentage of treatment discontinuation or interruptions | Baseline to Month 15
  Proportion of treatment discontinuation or interruptions for safety/ tolerability reason

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (37):
- France (13):
  - Novartis Investigative Site, Bayonne, Bayonne Cedex
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Gonesse
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Poissy
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Strasbourg
- Germany (10):
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Westerstede Olden
- Italy (5):
  - Novartis Investigative Site, Montichiari, BS
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Napoli
- Spain (9):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Salt, Girona
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com